CLINICAL TRIAL: NCT03094364
Title: Video Game-based Therapy for Arm Weakness In Progressive Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Lowell (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Lynne Gauthier, Associate Professor of Physical Therapy and Kinesiology, University of Massachusetts, Lowell
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60052127
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Primary Progressive Multiple Sclerosis; Hemiparesis
Keywords: Constraint-induced movement therapy; video game; virtual reality; upper extremity; CI therapy; rehabilitation; hemiparesis; MS; multiple sclerosis; progressive multiple sclerosis; primary progressive multiple sclerosis; secondary progressive multiple sclerosis; motor; physical therapy; physiotherapy; occupational therapy; arm; hand
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Paresis; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Treatment (Active Comparator): Patients will receive an in-home consultation with an occupational/physical therapist in which they are educated about the intervention, the system is set up, and they are guided through use of the system. After initial contact, therapist support will be available via telephone to address specific difficulties with operating the system, as well as three additional home visits throughout the 3 week intervention.
  The rehabilitation program requires use of the rehabilitation gaming system for 1.5 hours daily for 21 consecutive days (equivalent dosage to standard CI therapy), limb activation device worn for 90% of waking hours, and completion of the automated transfer package to facilitate real-world arm use (e.g., problem-solving modules, daily monitoring of arm use). After completing the intervention, the patient will receive additional consultation with the therapist to formulate goals for follow-up. Follow-up assessments will be conducted to assess long-term retention of motor gains.
  Interventions: Behavioral: Gaming CI Therapy
- Delayed Treatment (Active Comparator): Patients will receive an in-home consultation with an occupational/physical therapist in which they are educated about the intervention, the system is set up, and they are guided through use of the system. After initial contact, therapist support will be available via telephone to address specific difficulties with operating the system, as well as three additional home visits throughout the 3 week intervention.
  The rehabilitation program requires use of the rehabilitation gaming system for 1.5 hours daily for 21 consecutive days (equivalent dosage to standard CI therapy), limb activation device worn for 90% of waking hours, and completion of the automated transfer package to facilitate real-world arm use (e.g., problem-solving modules, daily monitoring of arm use). After completing the intervention, the patient will receive additional consultation with the therapist to formulate goals for follow-up. Follow-up assessments will be conducted to assess long-term retention of motor gains.
  Interventions: Behavioral: Gaming CI Therapy

INTERVENTIONS:
Behavioral: Gaming CI Therapy — Intensive remote (via video game) therapy for upper extremity hemiparesis.

SUMMARY:
Participants will receive intensive therapy through a video game in their own homes for 1 month. The game is operated by movements of the body (no controller needed) and acts like a virtual therapist. Participants will agree to play the game for 30 hours. They will also receive 4 home visits from a therapist designed to increase use of their arm for daily activities that are important to them. Participants will also receive a smart watch that will measure use of their weaker arm and alert them when their arm is not participating in activities. Arm strength and function will be measured before and after the therapy program.

DETAILED DESCRIPTION:
Randomized waitlist control trial. One group will receive treatment immediately (50%) and the other group will receive treatment following a three-week delay (50%). Group 1 will be assessed by physical/occupational therapists and rehabilitation psychologists (blinded to treatment phase) before and after the virtual gaming treatment. Group 2 will receive two baseline assessments (baseline followed by three weeks of usual and customary care and then another baseline before starting the gaming treatment), and again after three weeks of virtual gaming treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have progressive multiple sclerosis resulting in upper extremity motor impairment.
* Have the ability to comprehend and participate in basic elements of the therapy.
* Have substantial non-use in the more affected upper extremity.

Exclusion Criteria:

* Are currently participating in other experimental trials.
* Are currently participating in additional upper extremity therapy.
* Experienced relapse within the past 6 months.
* Too frail to undergo intensive rehabilitation,
* Those with serious, uncontrolled medical problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-11; Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Bilateral Activity Monitors (Accelerometers) | 0 to 1 Months
  Devices to monitor upper extremity movement throughout treatment
Wolf Motor Function Test | 0 to 1 Months
  Assessment to evaluate motor function

SECONDARY OUTCOMES:
Biomechanical Measures | 0 to 1 Months
  Recorded during game play through limb activation device and Kinect
Multiple Sclerosis Impact Scale (MSIS-29) | 0 to 1 Months
  Scale to asses living with MS
Short form-36 Health Survey | 0 to 1 Months
  Survey
Neuro-QOL | 0 to 1 Months
  Assessment to measure quality of life
Patient Health Questionnaire (PHQ-9) | 0 to 1 Months
Montreal Cognitive Assessment (MoCA) | 0 to 1 Months
  Assessment to measure cognitive function

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, 2154 Dodd Hall, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made public 1 year after study completion.